CLINICAL TRIAL: NCT01625091
Title: Pharmacotherapy for Alcohol Consumption in HIV Infected Women: Randomized Trial
Brief Title: Clinical Trial to Reduce Drinking in Women With HIV
Acronym: WHATIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida International University (Other); University of Miami (Other); Rush University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 86-2012-N; U01AA020797-01 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2012-06-21 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: HIV Infection
Keywords: HIV; women; drinking; Naltrexone
MeSH Terms: conditions — HIV Infections | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- naltrexone (Active Comparator): The investigators will administer Naltrexone to women with hazardous drinking and assess the study outcomes.
  Interventions: Drug: Naltrexone
- placebo pill (Placebo Comparator): The investigators will administer an inert placebo that looks similar to Naltrexone, to women with hazardous drinking and assess the study outcomes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — The study involves taking the drug naltrexone for up to 4 months. This will be given in a single pill each day for 4 months.
  Arms: naltrexone
Drug: Placebo — Placebo is an inert pill that looks the same as naltrexone. The placebo will be taken once each day for up to 4 months.
  Arms: placebo pill

SUMMARY:
The primary objective of this study is to evaluate whether an intervention that involves the medication naltrexone, will reduce drinking and improve health outcomes in women with HIV infection and hazardous drinking. Our central hypotheses are that, compared to women who receive placebo (sugar pill containing no medicine), women who receive naltrexone will have decreased rates of hazardous drinking, improved HIV medication adherence, less rapid disease progression, and reduced sexual risk behavior. The study design will involve 240 HIV-infected women with hazardous drinking, who will be recruited from HIV clinics, neighborhoods and referrals in Miami, Florida.

Eligible women will receive either a daily pill containing naltrexone (50mg) or an identical-appearing placebo for four months. All participants will receive encouragement and feedback related to their drinking regardless of medication assignment. The study participants will be assessed at two, four and seven months after enrollment. The proposed work is innovative because pharmacologic treatment for alcohol has not been evaluated in HIV-infected women. If our hypotheses are confirmed, the study findings would transform the approach to hazardous drinking within clinics serving HIV-infected women.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the acceptability and effectiveness of a treatment program for hazardous drinking, delivered within HIV-clinic outpatient settings, that involves oral naltrexone. The central hypothesis is that women participating in the treatment program will have decreased rates of hazardous drinking and improved clinical and behavioral health outcomes that are associated with hazardous drinking. The investigators have formulated this hypotheses based on the existing literature, the preliminary data and the clinical experience. The investigators theorize that women who receive an alcohol treatment intervention will be less likely to have "at risk" drinking behavior 6-months after enrollment, compared to women who received similar assessments but no formal treatment intervention. The investigators hypothesize that 4-months after enrollment, women who receive an alcohol treatment intervention will have improved adherence to HIV antiretroviral therapy, improved CD4 cell counts, reduced HIV viral load, and reduced risky sexual behavior, compared to women who receive similar assessments but no formal intervention.

The investigators will recruit 240 women from one site in Miami, Florida. Of those 240 women 120 will receive naltrexone and the others will receive placebo. Study participants will take the medication for 4 months but the investigators will follow them for 7 months. At baseline, 2 months, 4 months and 7 months, the investigators will administer study questionnaires and assess their liver enzymes, CD4 count and viral load. The investigators will also follow them up at months 1 and 3 to reinforce the medication intake and to assess for any possible side effects.

New treatment options are available, but their impact on hazardous drinking has not yet been evaluated among HIV-infected women, many of whom are poor, minorities, or who have associated mental health or substance abuse problems. Delivery of therapeutic interventions must be improved in order to reduce hazardous drinking in women with HIV/AIDS. The proposed research is significant because the therapy will be offered within HIV clinic settings and will potentially improve the health of a population that is significantly undertreated. In addition to determining the effectiveness of an alcohol treatment intervention, the investigators will also identify key barriers and facilitators associated with adherence to pharmacologic treatment for alcohol in women with hazardous drinking. The findings will directly affect the type and quality of care for hazardous drinking in this subset of HIV-infected individuals and will inform both primary and secondary prevention efforts.

ELIGIBILITY:
Inclusion Criteria: (must meet all of following):

* Hazardous drinking, on average, during the preceding 4 weeks. Defined as binge drinking (4 or more drinks per occasion at least twice monthly) and/or high total weekly consumption (>7 drinks per week).
* Age 18 or over
* Female
* HIV infection (documented by medical record blood test result or testing done for this study)
* Able to understand and comply with study procedures and to provide written consent.

Exclusion criteria: (cannot have any of the following):

* Contraindications to treatment with naltrexone
* Current physiologic opiate dependence
* Current daily prescription opioid medications
* Positive urine drug test for opioids
* Allergic to naltrexone
* Significantly abnormal baseline liver enzymes (AST or ALT >=5 times upper normal), evidence of acute hepatitis, or receiving hemodialysis for renal failure
* Currently pregnant
* Currently taking an alcohol treatment medication (disulfiram, topiramate, naltrexone, acamprosate).
* Currently unable to provide mailing address or reliable contact information, or has plans to move from area within next 7 months
* Unable to communicate in English or Spanish
* Research coordinator assessment that participant cannot comprehend the study or consent procedures (e.g. participant appears to be intoxicated, answers questions in a non-sensible manner)
* Has current prognosis of less than one year to live (e.g. in Hospice, has metastatic cancer)
* Currently taking antiviral treatment for hepatitis C infection (interferon or ribavirin)
* Has other unique health condition, not specifically listed, that should exclude the participant after discussion with Dr. Cook, Dr. Espinoza, and perhaps also the participant's primary HIV physician (for example an unexpected abnormal laboratory result turns up on the baseline screening metabolic panel).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Cook, MD, MPH, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Miami, Coral Gables, Florida
  - Florida International University, Miami, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: The participants took the drug naltrexone one single pill (50mg) each day for up to 4 months and then received final assessment at 7-months.
- Placebo: The participants took an inert placebo one single pill each day for up to 4-months and then received final assessment at 7-months. Placebo is an inert pill that looks the same as naltrexone.
Period: Intervention
Arm/Group | Naltrexone | Placebo
Started | 96 | 98
2 Months | 90 | 93
4 Months | 85 | 87
Completed | 85 | 87
Not Completed | 11 | 11
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 4 | 4
Not completed — Study termination | 2 | 3
Period: Post-intervention
Arm/Group | Naltrexone | Placebo
Started | 85 | 87
7 Months | 81 | 85
Completed | 81 | 85
Not Completed | 4 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Study termination | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (8.5) | 48.9 (8.9) | 48.3 (8.7)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-39 | 16 | 13 | 29
  Age group: 40-49 | 35 | 32 | 67
  Age group: 50-59 | 37 | 43 | 80
  Age group: ≥60 | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 98 | 194
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 11 | 11 | 22
  Race/Ethnicity: Not Hispanic, White | 3 | 5 | 8
  Race/Ethnicity: Not Hispanic, Black | 81 | 80 | 161
  Race/Ethnicity: Not Hispanic, Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Quit Hazardous Drinking
Description: The primary statistical outcome for the trial is alcohol consumption at month 4 when the drug is stopped. This main outcome is a categorical variable of either quit hazardous drinking (defined as ≤7 drinks per week and <4 drinks on any single day in the past 30 days), or did not quit (drinking exceeds the hazardous amount) .
Time Frame: Month 4
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 85 | 87
Participants | 44 | 39
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.36, Chi-squared

2. Secondary Outcome: Number of Binge Drinking Days
Description: In the past 30 days, total number of days with binge drinking which was defined as consuming ≥4 drinks on a single day (measured by Timeline Follow Back).
Time Frame: Month 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 85 | 87
Days | 0 [0 to 1] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Drinking Problems (SIP-2R Score)
Description: The Short Inventory of Problems (SIP-2R) seeks to measure the consequences of drinking in participants through questions related to guilt, reliability etc. The SIP-2R has 15 items asking how often the event happened during the past 3 months. Each item has a score from 0-3 (0=Never, 1=once or a few times, 2=once or twice a week, 3=daily or almost daily). The 15 questions from the SIP-2R are summed to create a total range of scores from 0-45.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 85 | 87
units on a scale | 7.2 (9.9) | 6.7 (8.4)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.70, t-test, 2 sided

4. Secondary Outcome: Craving for Alcohol
Description: Self-reported scale of alcohol craving ranging from 0 (no craving) to 10 (strongest craving)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 85 | 87
units on a scale | 3.3 (3.4) | 3.2 (2.9)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.98, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/96 | 2/98
Serious Adverse Events (participants affected / at risk) | 10/96 | 6/98
Other Adverse Events (participants affected / at risk) | 77/96 | 74/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=96) | Placebo (N=98)
Inpatient hospitalization (General disorders) | 10 (10) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=96) | Placebo (N=98)
Nausea (Gastrointestinal disorders) | 35 | 29
Diarrhea (Gastrointestinal disorders) | 23 | 27
Headache (Nervous system disorders) | 28 | 19
Fatigue (General disorders) | 28 | 18
Decreased appetite (General disorders) | 21 | 23
Depression (Psychiatric disorders) | 27 | 16
Sleepiness (General disorders) | 24 | 19
Dizziness (General disorders) | 23 | 14
Itchiness (Skin and subcutaneous tissue disorders) | 15 | 21
Nervousness/Anxiety (Psychiatric disorders) | 16 | 18
Abdominal pain (General disorders) | 20 | 13
Vomiting (Gastrointestinal disorders) | 22 | 8
Insomnia (General disorders) | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No